CLINICAL TRIAL: NCT06937541
Title: Family Interventions iN Dementia Mental Health Environments
Acronym: FIND ME
Status: Recruiting | Type: Observational
Sponsor: University of West London (Other)
Collaborators: University of Cambridge (Other); University of Exeter (Other)
Responsible Party: Principal Investigator, Emma Wolverson, Professor, University of West London
Other Study IDs: NIHR161439; NIHR161439 (Other Grant/Funding Number: National Institute of Health Research (NIHR))
Record Dates: First submitted 2025-03-21; First posted 2025-04-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Carers; Dementia
Keywords: family carers; dementia; inpatient unit; mental health; family interventions
MeSH Terms: conditions — Dementia; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Ward managers of dementia mental health wards: Ward managers of mental health wards that provide specialist care to patients with dementia will be invited to participate in a UK-wide, national mapping survey. One ward manager per ward is required to complete survey. Ward managers from NHS trusts and private providers will be invited to participate. There are approximately 90 NHS wards and 20 private providers in the UK (e.g. Cygnet Health Care, the Priory Group, Elysium Health Care, and St Andrew's Healthcare). Target recruitment goal of survey completion is 50% = 55 ward managers in total.
- Co-design study participants: Co-design workshops will be conducted with people living with dementia (n=10) and carers (n=10), and staff (n=10) working on mental health wards, to translate the findings into evidence-based strategies and collaboratively shape service improvements to address user needs and enhance care.
- Feasibility study participants: People living with dementia (n=30), carers (n=30) and staff (n=30) will be recruited to test the feasibility of resources and interventions, co-designed to improve carer support, involvement and staff training.
- Family carers: Interviews will be conducted with family carers whose friend/relative has received care on a dementia mental health ward (recruitment will take place across 3 wards). The investigators will interview current carers (8 per ward, total = 24) at 3 time points over 1 year. They will be carers of patients with dementia currently receiving care on a mental health ward. The investigators will also interview carers whose friend/relative has been discharged from a mental health ward within the last 3 years (8 per ward, total = 24).
  People with dementia receiving care on mental health wards are usually in the advanced stages of dementia and very distressed. However, there may be some who have the capacity to consent and if they wish, will be supported in taking part in dyadic interviews with their carer.
- Health care professionals working on a dementia mental health ward: Ethnographic observations will be conducted of staff working on dementia mental health wards. These will be focused on how staff interact with, support and involve family carers in the decisions of the care of their friend/relative with dementia receiving care on the ward.
  In-situ ethnographic interviews (5-10 mins reciprocal conversations) with ward staff will take place during observations to explore what staff draw on to inform their interactions and support with carers, how they recognise carers needs and what informal and embedded rationales used in decision making inform their involvement with carers.
  Staff to take part in longer (30-60 min) interviews (5 per site, total = 15) will be identified in collaboration with ward managers. The sample will include staff from a range of disciplines and roles.

SUMMARY:
Study Goal: Understand carers' needs when someone with dementia is in a mental health ward and develop strategies to support carers as partners in care.

Research Questions:

* What are mental health wards like in terms of staff, patients, and current carer support?
* What do carers experience and need during admission, discharge, and beyond?
* How do ward routines and staff practices affect carer involvement?
* How can co-design turn research into practical strategies for carer support?
* Can these strategies be implemented effectively?

Method: The investigators will survey mental health wards nationwide, interview carers from three UK wards, observe ward practices, and talk to staff. They will use this information to create and share practical strategies to improve carer support across the UK.

DETAILED DESCRIPTION:
Background and rationale

Mental health wards (MHW) are a significant site of care for people living with dementia (PLWD), providing care for the most unwell, vulnerable, and high-risk individuals who are detained under the Mental Health Act (1983) for their own safety and the safety of others.

The UK has around 100 MHWs (80 NHS, 20 private) for PLWD, but there's a lack of evidence on care quality and experiences. Stays average 100 days, with most PLWD moving to institutional care rather than returning home.

Admissions often follow severe psychiatric or behavioural issues, such as self-harm or assaults. This population is at high risk to themselves and others, with high acuity and comorbidity. Admissions are complex, involving frequent unscheduled transfers to general hospitals, which are associated with high rates of falls and hospital-acquired infections.

Carer involvement can significantly improve clinical and social outcomes for people in mental health wards by reducing length of stay, promoting earlier discharge, and lowering relapse and readmission rates. Carers provide essential support that staff may not, ensuring person-centred care, advocacy, decision-making support, treatment adherence, and promoting recovery. However, carers often feel marginalized and describe MHWs as a place of 'battle,' experiencing high levels of trauma and distress with unmet emotional, social, and financial needs. Reviews and inquires highlight a culture that views carers as problematic and resource-intensive, leading to their support needs being overlooked.

There is an absence of research examining carer perspectives of MHWs and no evidence-based interventions to support carers of PLWD who are admitted within MHWs. In response, this study responds to urgent calls from the Department of Health and Social Care and NHS England, for partnership working with carers and families utilising co-production to develop effective interventions and training programmes to support carers and the guidance required by services and wards to support implementation.

Research question: How can MHWs effectively work in partnership with and support family carers of PLWD?

Aim and Objectives

This study will provide detailed understandings of carers experiences and involvement when PLWD are detained within a MHW, and staff rationales and responses to carers, throughout an admission. It will deliver new knowledge and evidence-based strategies co-designed to ensure carers are appropriately supported and involved and to improve patient outcomes.

Objectives:

1. To deliver a detailed description of staffing structure, patient profiles, and current support for carers and families in MHWs for PLWD.
2. Provide detailed understandings of carers' experiences, perspectives of involvement, and their support needs throughout a PLWD MHW admission, during transition, and following discharge.
3. Understand ward organisational cultures and staff perspectives by examining (a) ward routines and practices that involve or exclude carers (b) staff understandings and recognition of carers needs, and (c) formal frameworks and informal rationales staff draw on to inform involvement or exclusion from decision making, care, and transition to discharge.
4. Translate the findings using co-design into evidence-based strategies to support best practice in the involvement and support of carers.
5. (a) Assess the feasibility of implementing these strategies in practice and (b) gather feedback from people with lived experience

Design

This mixed methods study uses a convergent parallel mixed methods design integrating a national mapping survey, interviews, ethnography and experience-based co-design and feasibility testing. This approach supports the collection of detailed data from multiple and contextualized perspectives, with the goal to improve healthcare systems.

The study uses family systems theory and the Family Adjustment and Adaptation Response Model (FARR) to understand family responses to stress, such as dementia and mental health admissions. It also incorporates anthropology and sociology theories to explore family and kinship in care contexts and how healthcare professionals and MHWs recognize and respond to families. This combined approach aims to understand carers' and families' experiences and how to best support them during MHW admissions.

ELIGIBILITY:
Survey

Inclusion Criteria:

* Ward managers of mental health wards that provides care to PLWD
* Ward managers from NHS wards that provides care to PLWD
* Ward managers from private providers that provides care to PLWD
* Ward managers that work on organic or mixed wards that provides care to PLWD

Exclusion Criteria:

* Functional older adult mental health wards that do not provide care to PLWD
* Staff members who are not the ward manager

Longitudinal interviews with current carers

Inclusion criteria:

* Family member (any relationship) or friend of a PLWD currently receiving care on a mental health ward
* Aged 18 years old or above
* Has capacity to consent to participate in an interview
* Willing to take part in 3 interviews over 12 months

Exclusion criteria:

* The carer is actively involved in a safeguarding investigation.
* The carer is under 18 years old
* The carer does not have capacity to consent to participate in an interview

Interviews with discharged carers

Inclusion criteria:

* Family member (any relationship) or friend of a PLWD discharged from the ward within the last 3 years
* Aged 18 years old or above
* Has capacity to consent to participate in an interview
* Willing to take part in an interview

Exclusion criteria:

* The carer is actively involved in a safeguarding investigation
* The carer is under 18 years old
* The carer does not have capacity to consent to participate in an interview

Interviews with People Living With Dementia (PLWD)

Inclusion criteria:

* PLWD currently under the care of the mental health ward
* PLWD discharged from the care of a dementia mental health ward within the last 3 years
* Has capacity to give informed consent to taking part in an interview
* Willing to take part in an interview alongside their carer

Exclusion criteria:

* The PLWD is actively involved in a safeguarding investigation
* The PLWD does not have capacity to consent to participate in an interview
* The PLWD is not willing to take part in an interview alongside their carer
* The PLWD has been discharged from the care of a dementia mental health ward for more than 3 years

Co-design study - PLWD and carers

Inclusion criteria:

* PLWD who may, or may not, have experience of dementia mental health wards
* Carers (family members or friends) of PLWD who may, or may not, have experience of dementia mental health wards
* Willing to talk about mental health and dementia
* Aged 18 years old or above
* Have capacity to give informed consent

Exclusion criteria:

* Participants who do not have experience of living with, or caring for someone with, dementia
* Not willing to talk about mental health and dementia
* Aged under 18 years old
* Does not have capacity to give informed consent

Co-design study - staff

Inclusion criteria:

* Members of staff working within mental health wards for PLWD
* Members of staff of any professional group in a role that involves contact with carers (e.g. health care assistants, nurses, occupational therapists, psychologists, physiotherapists, speech and language therapists, family therapists, psychiatrists etc)
* Members of staff of any pay band or grade
* Students on placement in a mental health ward
* Members of staff working on NHS or private wards

Exclusion criteria:

* The staff member is actively involved in a safeguarding investigation
* Members of staff that do not work within mental health wards for PLWD

Feasibility study - PLWD and carers

Inclusion criteria:

* PLWD
* Carer (family or friend; current or bereaved)
* Willing to review outputs related to mental health wards
* Aged 18 years old or above
* Capacity to consent to take part

Exclusion criteria:

* The participant (PLWD or carer) is actively involved in a safeguarding investigation.
* Is not willing to review outputs related to mental health wards
* Aged under 18 years old
* Does not have capacity to consent to take part

Feasibility study - staff

Inclusion criteria:

* Members of staff working within mental health wards for PLWD
* Members of staff of any professional group in a role that involves contact with carers (e.g. health care assistants, nurses, occupational therapists, psychologists, physiotherapists, speech and language therapists, family therapists, psychiatrists etc)
* Members of staff of any pay band or grade
* Students on placement in a mental health ward
* Members of staff working on NHS or private wards

Exclusion criteria:

* The staff member is actively involved in a safeguarding investigation
* Members of staff that do not work within mental health wards for PLWD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People living with dementia, their carers and staff working on the mental health wards
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
A national survey to map current care provision for people living with dementia admitted to a mental health ward across the UK | 6 months
  National mapping survey to gather data on the number/type of wards, patient and staff demographics and existing care provision for people living with dementia who are detained under the Mental Health Act and receiving care on a mental health ward.
Ethnographic observations to understand how carers are supported and involved in the care of their friend/relative with dementia receiving care on a mental health ward | 1 year
  Ethnographic observation of staff and family carers on the ward. The focus of the observations is on the organisation of care. Observations will take place from the corridor(s) of wards, in communal areas, typically at nursing stations or ward observation points. Short, 'in-situ' conversational interviews (around 5-10 minutes) will take place on the ward with staff. These will be unstructured conversations to capture 'in-the-moment' experiences. Observations and 'in-situ' conversations will be documented using a touch screen tablet device.
Interviews with current carers to understand their experiences and involvement in the care of their friend/relative with dementia who is receiving care on a mental health ward | 1 year
  Interviews with carers across 3 NHS sites in the UK, who currently have a friend/relative with dementia receiving care on a mental health ward (8 carers per ward = 24 carers in total). Carers will be interviewed at 3 timepoints over 12 months to understand their experiences over time. Total number of interviews = 72. The sample of carers will be identified by ward managers. A semi-structured interview schedule will be used following a narrative interview approach.
Interviews with discharged carers to understand their experiences and involvement in the care of their friend/relative with dementia who had previously received care on a mental health ward | 1 year
  Interviews with 'discharged' carers across 3 NHS sites, i.e. carers whose friend/relative with dementia had previously received care on a mental health ward and have been discharged from the ward within the last 3 years. 8 carers per ward = 24 interviews in total. The sample of carers will be identified via screening of ward records completed by ward managers at each ward. A letter and Participant Information Sheet (PIS) will be sent by post to invite discharged carers to participate in an interview. A semi-structured interview schedule will be used to capture their views and experiences.
Interviews with ward staff to understand their experiences of supporting and involving carers in the care of their friend/relative with dementia receiving care on a mental health ward | 1 year
  Interviews with ward staff, such as nurses, healthcare assistants, psychiatrists across 3 NHS sites. 5 ward staff per site will be interviewed = 15 interviews. Ward staff will be identified in collaboration with ward managers. A semi-structured interview schedule will be used to capture their views and experiences.
Focus groups with staff to assess the feasibility (acceptability, implementation, integration, relevance) of implementing co-designed strategies in practice | 6 months
  Focus groups with staff to address:
  i) acceptability, to what extent these strategies reflect current practice, constraints, and the potential for new approaches; ii) implementation, to what extent they can be successfully delivered; iii) integration, to what extent they can be integrated into routine practice iv) relevance and acceptability of the outputs created for PLWD, carers and families.
  Three online focus groups of 8-10 participants (n=30) will provide opportunity for discussion to explore the structural and organisational barriers within wards that may facilitate or impede effective implementation.
Acceptability of co-designed strategies and resources | 6 months
  PLWD, carers and families will be invited to share their perspectives around acceptability of the co-designed resources in a way that suits them most. This is a person-centered, inclusive approach to gathering feedback, where different approaches are paramount to suit different needs.
  People with lived experience could share their feedback by annotating printed or electronic versions of documents, having a brief conversation with the researcher online, over the phone or in person via the researcher attending their PPI meetings.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Emma Wolverson, DClinPsy, Principal Investigator — University of West London
Locations (1):
- Geller Institute of Aging and Memory, University of West London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD which underlie results in any publications will be shared and made available on an online repository. No identifiable patient data will be shared; all data will be anonymised.

REFERENCES:
- [Background] Edmans BG, Wolverson E, Dunning R, Slann M, Russell G, Crowther G, Hall D, Yates R, Albert M, Underwood BR. Inpatient psychiatric care for patients with dementia at four sites in the United Kingdom. Int J Geriatr Psychiatry. 2022 Feb;37(2). doi: 10.1002/gps.5658. Epub 2021 Dec 1. No abstract available. PMID 34850970
- [Background] Wolverson EL, Harrison Dening K, Dunning R, Crowther G, Russell G, Underwood BR. Family experiences of inpatient mental health care for people with dementia. Front Psychiatry. 2023 Mar 1;14:1093894. doi: 10.3389/fpsyt.2023.1093894. eCollection 2023. PMID 36937714
- [Background] Wolverson E, Dunning R, Crowther G, Russell G, Underwood BR. The Characteristics and Outcomes of People with Dementia in Inpatient Mental Health Care: A Review. Clin Gerontol. 2024 Oct-Dec;47(5):684-703. doi: 10.1080/07317115.2022.2104145. Epub 2022 Jul 27. PMID 35897148
- See also: URl for the FIND ME Study Website — https://www.uwl.ac.uk/research/research-centres-and-groups/geller-institute-ageing-and-memory/research/findme